CLINICAL TRIAL: NCT03177707
Title: Mindfulness-based Therapy Group Intervention for Couple's Dealing With Sexual Dysfunction After Prostate-cancer Treatment
Brief Title: Intimacy and Mindfulness Post-Prostate Cancer Treatment
Acronym: IMPPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vancouver Prostate Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IMPPACT
Record Dates: First submitted 2017-03-07; First posted 2017-06-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer; Sexual Dysfunction
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological | interventions — Family Characteristics

STUDY DESIGN:
Intervention Model Description: Couples will be randomized to an immediate or delayed treatment group; the delayed treatment couples will be considered the waitlist control group in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate start (Experimental): Patients begin the Mindfulness-based Therapy Group for Couples treatment group immediately after enrollment
  Interventions: Other: Mindfulness-based Therapy Group for Couples
- Delayed start (Other): Patients begin the Mindfulness-based Therapy Group for Couples after a delay post-study enrollment (approximately 6 months)
  Interventions: Other: Mindfulness-based Therapy Group for Couples

INTERVENTIONS:
Other: Mindfulness-based Therapy Group for Couples — Eligible couples will take part in a 4-session mindfulness-based therapy group for couples. The groups will last 2 hours in length, for a total of 8 hours of treatment time, and sessions will be scheduled once per week in successive weeks.
  The groups will have one highly experienced female facilitator, who is the Study Coordinator. The facilitator led the design of the treatment manual, and has experience in facilitating similar groups. The facilitator will follow a detailed, empirically-informed mindfulness-based treatment manual that was designed for the purpose of this study. All groups will take place in a private group treatment room at Vancouver General Hospital.

SUMMARY:
With improvements in detection and treatment of prostate cancer (PCa), more men than ever are living with side effects from PCa treatment; most distressingly, treatment side effects include problems with sexual functioning (e.g. erectile dysfunction, climacturia, inorgasmia). This study aims to develop a mindfulness-based group treatment for couples with sexual functioning complaints post-PCa treatment. Couples will be invited to a four-session mindfulness-based treatment group. Pre- and post-treatment outcomes (e.g., distress, sexual functioning/enjoyment, relationship satisfaction, treatment adherence) will assess feasibility and effectiveness of this novel treatment for couple's sexual lives after PCa.

DETAILED DESCRIPTION:
This is an intervention study designed to assess a novel mindfulness-based treatment protocol for couples dealing with sexual dysfunction secondary to prostate cancer treatment. Couples will be invited to participate through the Vancouver Prostate Centre (VPC) and the Prostate Cancer Survivorship Care (PCSC) Program. Interested couples will be screened for eligibility. Eligible couples will be randomized to either an immediate-start or a delayed-waitlist control group.

Prior to treatment, couples will complete an online questionnaire package. Treatment will consist of a 4-week mindfulness-based group lead by a clinician trained in mindfulness treatment. Sessions are 2hrs in length and take place in consecutive weeks, with daily homework recommended between sessions. The intervention was developed based on pre-existing mindfulness-based cognitive therapy treatment groups for sexual dysfunction developed by Dr. Lori Brotto at the UBC Sexual Health Laboratory, mindfulness in sex therapy and intimate relationships (MSIR) treatment group developed by Kocsis and Newbury-Helps (2016), and expert input. Sessions consist of mindfulness-based training, sex therapy techniques, and education. After treatment, couples will be invited to complete a post-treatment questionnaire once immediately after the end of treatment, and again 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a relationship that has lasted longer than 1 year
* Both members of the couple are at least 19 years of age or older
* Both members of the couple are able to speak and read English (to date, all of the treatment material is delivered in English)
* (At least) one member of the couple has a history of prostate cancer diagnosis
* The same member of the couple underwent radical prostatectomy for the treatment of his prostate cancer
* Both members of the couple are willing and able to comply with all study procedures (including committing to daily homework over the 4-week period of the treatment program) and be available for the duration of the study
* Both members of the couple provide signed and dated informed consent form

Exclusion Criteria:

* The individual who was treated with prostate cancer received androgen deprivation therapy or radiation therapy to treat their prostate cancer.
* Have a current health condition (e.g., severe cardiovascular health problems, unmanaged diabetes mellitus), physical disabilities, or mental health issues (e.g., severe anxiety, depression) that would interfere with self- or partnered-sexual activities, or the individual's ability to attend group sessions or complete home assignments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Sexual correlates: Self-reported sexual functioning | Change from baseline to post-intervention (5 weeks)
  Depending on sexual orientation and gender, individuals will complete either (1) International Index of Erectile Functioning (heterosexual men), International Index of Erectile Functioning for Men who have sex with men (gay men), or Female Sexual Functioning Index (female partners)
Sexual correlates: Self-reported erectile functioning | Change from post-intervention (5 weeks) to 6-month follow up
  Depending on sexual orientation and gender, individuals will complete either (1) International Index of Erectile Functioning (heterosexual men), International Index of Erectile Functioning for Men who have sex with men (gay men), or Female Sexual Functioning Index (female partners)
Sexual correlates: GMSEX | Change from baseline to post-intervention (5 weeks)
  GMSEX (Lawrance & Byers, 1992). The GMSEX is a 5-item measure of distress related to sexual functioning with one's partner.
Sexual correlates: GMSEX | Change from post-intervention (5 weeks) to 6-month follow up
  GMSEX (Lawrance & Byers, 1992). The GMSEX is a 5-item measure of distress related to sexual functioning with one's partner.
Sexual correlates: Sexual activity scale | Change from baseline to post-intervention (5 weeks)
  This is a questionnaire developed by the study lead that asks individual to rate the frequency of times that they engaged in a range of sexual activities over 3 time-periods: (a) ever, (b) since their/their partner's prostate cancer surgery, and (c) in the past 4 weeks.
Sexual correlates: Sexual activity scale | Change from post-intervention (5 weeks) to 6-month follow up
  This is a questionnaire developed by the study lead that asks individual to rate the frequency of times that they engaged in a range of sexual activities over 3 time-periods: (a) ever, (b) since their/their partner's prostate cancer surgery, and (c) in the past 4 weeks.
Sexual correlates: Adapted dyadic adjustment scale | Change from baseline to post-intervention (5 weeks)
  Adapted dyadic adjustment scale (A-DAS; Sharpley & Cross, 1982). The A-DAS is a validated, 7-item measure that assesses relationship adjustment.
Sexual correlates: Adapted dyadic adjustment scale | Change from post-intervention (5 weeks) to 6-month follow up
  Adapted dyadic adjustment scale (A-DAS; Sharpley & Cross, 1982). The A-DAS is a validated, 7-item measure that assesses relationship adjustment.

SECONDARY OUTCOMES:
mental and health-related quality of life indices: Hospital Anxiety and Depression Scale | Change from baseline to post-intervention (5 weeks)
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983). The HADS is a validated, 14-item measure of depression and anxiety..
mental and health-related quality of life indices: Hospital Anxiety and Depression Scale | Change from post-intervention (5 weeks) to 6-month follow up
  Hospital Anxiety and Depression Scale (HADS; Zigmond & Snaith, 1983). The HADS is a validated, 14-item measure of depression and anxiety..
mental and health-related quality of life indices: UCLA Prostate Cancer Index | Change from baseline to post-intervention (5 weeks)
  UCLA Prostate Cancer Index (Litwin, Hays, Fink, Ganz, Leake, & Brook, 1998). This is a 20-item measure that assesses health-related quality of life indices specific to common side effects of prostate cancer treatment.
mental and health-related quality of life indices: UCLA Prostate Cancer Index | Change from post-intervention (5 weeks) to 6-month follow up
  UCLA Prostate Cancer Index (Litwin, Hays, Fink, Ganz, Leake, & Brook, 1998). This is a 20-item measure that assesses health-related quality of life indices specific to common side effects of prostate cancer treatment.

OTHER OUTCOMES:
Treatment mechanisms factors: Five Facets of Mindfulness questionnaire Short form | Change from baseline to post-intervention (5 weeks)
  Five Facets of Mindfulness questionnaire; Short form (Bohlmeijer, E., P. M. ten Klooster, et al., 2011), which is a validated, 24-item measure of different aspects of attentiveness.
Treatment mechanisms factors: Five Facets of Mindfulness questionnaire Short form | Change from post-intervention (5 weeks) to 6-month follow up
  Five Facets of Mindfulness questionnaire; Short form (Bohlmeijer, E., P. M. ten Klooster, et al., 2011), which is a validated, 24-item measure of different aspects of attentiveness.
Treatment mechanisms factors: Expectations for treatment | Change from baseline to post-intervention (5 weeks)
  Expectations for treatment. A 4-item questionnaire, designed for and used in our approved mindfulness-based treatment study for women with provoked vestibulodynia
Treatment mechanisms factors: Expectations for treatment, | Change from post-intervention (5 weeks) to 6-month follow up
  Expectations for treatment. A 4-item questionnaire, designed for and used in our approved mindfulness-based treatment study for women with provoked vestibulodynia
Treatment mechanisms factors: Time since prostate cancer treatment | Change from baseline to post-intervention (5 weeks)
  This is a single-item, face-valid question asking participants to indicate time since prostate cancer treatment. Responses will be cross-validated by comparing against partner response and also information gathered from their chart, if they were recruited through the Sexual Health Service.
Treatment mechanisms factors: Time since prostate cancer treatment | Change from post-intervention (5 weeks) to 6-month follow up
  This is a single-item, face-valid question asking participants to indicate time since prostate cancer treatment. Responses will be cross-validated by comparing against partner response and also information gathered from their chart, if they were recruited through the Sexual Health Service.
Treatment mechanisms factors: Penile Rehabilitation Aids Use | Change from baseline to post-intervention (5 weeks)
  This questionnaire asks participants about their/their partner's use of penile rehabilitation aids, and their perception of these treatment usefulness will be asked.
Treatment mechanisms factors: Penile Rehabilitation Aids Use | Change from post-intervention (5 weeks) to 6-month follow up
  This questionnaire asks participants about their/their partner's use of penile rehabilitation aids, and their perception of these treatment usefulness will be asked.
Treatment mechanisms factors: Mindfulness Practice | Change from baseline to post-intervention (5 weeks)
  This is a questionnaire designed by the experimenters to assess the amount of daily mindfulness practice. Participants will indicate the number of minutes they spent practicing each day. This log will be completed as a separate, online questionnaire that participants will access daily. Participants have the option of completing a paper-version of this log, which they will give to the Study Coordinator each week.
Treatment mechanisms factors: Mindfulness Practice | Change from post-intervention (5 weeks) to 6-month follow up
  This is a questionnaire designed by the experimenters to assess the amount of daily mindfulness practice. Participants will indicate the number of minutes they spent practicing each day. This log will be completed as a separate, online questionnaire that participants will access daily. Participants have the option of completing a paper-version of this log, which they will give to the Study Coordinator each week.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No